CLINICAL TRIAL: NCT02455700
Title: A Hospital Based Prospective Randomised Controlled Clinical Trial Comparing Pain Experience Using Manual and Rotary Interproximal Enamel Reduction Techniques in Orthodontic Patients
Brief Title: Pain Associated With Interproximal Enamel Reduction in Orthodontics: a RCT
Acronym: IER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Niamh O'Rourke, Miss G Minhas, Consultant in Orthodontics, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IER V1 06.03.2015
Record Dates: First submitted 2015-05-20; First posted 2015-05-28 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Orthodontic, Interproximal Enamel Reduction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand driven enamel reduction (Active Comparator): This group will have enamel reduction in the lower incisor region carried out using hand held devices
  Interventions: Device: Interproximal Enamel Reduction
- Rotary ( motor driven) device (Active Comparator): This group will ahve enamel reduction in the lower incisor region carried out using a rotary (motor driven) device
  Interventions: Device: Interproximal Enamel Reduction

INTERVENTIONS:
Device: Interproximal Enamel Reduction — removal of enamel between lower incisor teeth as part of orthodontic treatment plan to achieve the aims of treatment
  Other Names: interdental stripping

SUMMARY:
Prospective randomised crossover trial to assess if there is a difference in the level of pain experienced by orthodontic patients undergoing interpromixal enamel reduction at the lower incisor region using either a motor driven reduction device or a hand held device

DETAILED DESCRIPTION:
Consenting participants will be randomly allocated to one of the two groups ( motor driven device or hand driven device). A pain questionnaire in the form of a Visual Analogue Scale will be used before the treatment to determine a baseline level of pain and after the chosen treatment to determine the effect or the intervention on pain experience.

After a washout period of 6 weeks the participants will crossover to have the opposite intervention carried out. A VAS will be filled in before and after the intervention again to determine a baseline pain score and pain score associated with the intervention.

The data will be gathered and entered electronically into a statistical package whereby appropriate statistics will be carried out to determine if there is a significant difference in pain experienced between the two methods of enamel reduction.

A secondary aim willl be to determine if there is any correlation with pain experienced and age or gender.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Requiring IER in the lower anterior teeth as part of treatment plan
* mild crowding in the lower incisor region
* centreline discrepancy
* discrepancy between the arches mild and thus requiring IPR to correct incisor position
* requiring IER for arch coordination No medications Willing to participate

Exclusion Criteria:

* Under 18 years of age Not requiring IER
* moderate or severe crowding necessitating extraction for relief of crowding
* patients with removable appliances as their only mode of treatment Patient taking medication Not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The level of pain associated with each type of enamel reduction technique will be measured using a 100mm visual analogue scale which will be filled out by participant | Two consecutive visits, 6 weeks apart, over a course of orthodontic treatment which usually lasts 18 to 24 months

SECONDARY OUTCOMES:
Level of pain experienced with respect to age and gender of participant as assessed by the visual analogue scale | Two consecutive visits, 6 weeks apart, over a course of orthodontic treatment which usually lasts 18 to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gursharan Minhas, MOrth, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (1):
- RSCH, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sudarshan S, Sherriff M, O'Rourke N, Minhas G. Difference in pain experience between manual and motor-driven methods of interproximal enamel reduction: a single centre randomized controlled trial. Eur J Orthod. 2025 Oct 16;47(6):cjaf074. doi: 10.1093/ejo/cjaf074. PMID 41229345